CLINICAL TRIAL: NCT01219842
Title: Invasive Revascularization or Not in Intermittent Claudication
Acronym: IRONIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Joakim Nordanstig, vascular surgeon, PhD student, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sahlgrenska Academy
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Intermittent Claudication
Keywords: Intermittent claudication; Health Related Quality of Life; Walking performance; Daily walking capacity
MeSH Terms: conditions — Intermittent Claudication | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- INVASIVE (INV) group (Active Comparator): Modern endovascular and/or open revascularization according to the recommendations in the TASC II document.
  Interventions: Procedure: INVASIVE (INV) treatment; Other: Best medical treatment (BMT)
- NON-INVASIVE (NON) group (Active Comparator): Patients receiving only best medical treatment (BMT).
  Interventions: Other: Best medical treatment (BMT)

INTERVENTIONS:
Procedure: INVASIVE (INV) treatment — Modern endovascular and/or open revascularisation according to the TASC II recommendations.
  Arms: INVASIVE (INV) group
Other: Best medical treatment (BMT) — Antiplatelet therapy, cilostazol and non-supervised exercise training. Smoking cessation support. Lipid-lowering therapy, diabetes and hypertension treated according to current national guidelines.

SUMMARY:
Peripheral arterial disease (PAD) often causes exertion pain in the legs, intermittent claudication (CI) affecting> 10% of individuals> 65 years. A recent Swedish Health Technology Assessment Report identified only limited evidence for the effectiveness of invasive treatment for IC in patients already on exercise training. The prognosis for the extremity is usually benign and treatment therefore aims at improving quality of life. Invasive treatment can also cause serious complications. Coronary artery disease is common in IC patients increasing the risk with invasive treatment. In spite of these uncertain merits and potential risks, invasive procedures for IC are increasing and 37% of all invasive procedures for PAD in Sweden are performed for IC. The aim of this study is to evaluate the additional effects of modern invasive treatment in patients with intermittent claudication receiving modern best medical treatment (BMT). The primary hypothesis in the study is that invasive treatment in addition to BMT improves health related quality of life and walking performance compared to BMT only.

ELIGIBILITY:
Inclusion Criteria:

* Patient with intermittent claudication (typical symptoms and ABI <0.9) seeking treatment
* Significant aortoiliac- and/or femoropopliteal lesion.
* Age 30-80 years

Exclusion Criteria:

* Invasive treatment contraindicated because of severe intercurrent disease.
* Two or more failed vascular reconstructions in the same leg.
* Employees unable to work because of intermittent claudication.
* Need for open reconstruction below the tibioperoneal trunc.
* Thromboembolic etiology (popliteal artery aneurysm; cardiac emboli)
* Other disease severely affecting walking performance.
* Body weight > 120 kilograms.
* Age <30 or > 80 years.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2010-03; Primary Completion 2014-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life (HRQOL) | 24 months with intermistic analysis at 12 months
  Assessed with the patient-reported instruments SF-36, EQ5D and VASCUQOL

SECONDARY OUTCOMES:
Walking performance on treadmill test | 24 months with interimistic analysis at 12 months
  Graded treadmill test with progressively increasing speed and inclination.
Health Related Quality of Life (HRQOL) | 60 months
  Assessed with the patient-reported instruments SF-36, EQ5D and VASCUQOL
Walking performance on treadmill test | 60 months
  Graded treadmill test with progressively increasing speed and inclination.
six-minutes walk test | 60 months
  Corridor-based walk test during six minutes walk

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Nordanstig, M D, Principal Investigator — Sahlgrenska Academy, Institute of Medicine, Department of Molecular and Clinical Medicine; Lennart Jivegård, M D, PhD, Study Director — Sahlgrenska Academy, Institute of Medicine, department of Molecular and Clinical Medicine; Klas Österberg, M D, PhD, Study Chair — Sahlgrenska Academy, Institute of Medicine, Department of Molecular and Clinical Medicine; Johan Millinger, MD, Study Chair — Sahlgrenska Academy, Institute of Medicine, Department of Molecular and Clinical Medicine
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Derived] Djerf H, Millinger J, Falkenberg M, Jivegard L, Svensson M, Nordanstig J. Absence of Long-Term Benefit of Revascularization in Patients With Intermittent Claudication: Five-Year Results From the IRONIC Randomized Controlled Trial. Circ Cardiovasc Interv. 2020 Jan;13(1):e008450. doi: 10.1161/CIRCINTERVENTIONS.119.008450. Epub 2020 Jan 15. PMID 31937137
- [Derived] Nordanstig J, Taft C, Hensater M, Perlander A, Osterberg K, Jivegard L. Two-year results from a randomized clinical trial of revascularization in patients with intermittent claudication. Br J Surg. 2016 Sep;103(10):1290-9. doi: 10.1002/bjs.10198. Epub 2016 May 25. PMID 27220310
- [Derived] Nordanstig J, Taft C, Hensater M, Perlander A, Osterberg K, Jivegard L. Improved quality of life after 1 year with an invasive versus a noninvasive treatment strategy in claudicants: one-year results of the Invasive Revascularization or Not in Intermittent Claudication (IRONIC) Trial. Circulation. 2014 Sep 16;130(12):939-47. doi: 10.1161/CIRCULATIONAHA.114.009867. Epub 2014 Aug 5. PMID 25095886